CLINICAL TRIAL: NCT04268914
Title: Effectiveness of Virtual Reality to Reduce Pre-Operative Anxiety
Brief Title: Virtual Reality to Reduce Pre-Operative Anxiety
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The AR technology we were using is now out of business and we are trying to use a different device.
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: AppliedVR Inc. (Industry)
Responsible Party: Principal Investigator, Jeffrey I Gold, PhD, Professor of Anesthesiology, Pediatrics, and Psychiatry & Behavioral Sciences, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHLA-15-00461
Record Dates: First submitted 2020-02-10; First posted 2020-02-13 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Virtual Reality; Augmented Reality; IV Stick; Mask Induction; Ambulatory Surgery; Pain; Anxiety
Keywords: virtual reality; augmented reality; IV stick; mask induction; tonsillectomy; adenoidectomy; arthroscopy; hernia; circumcision; orchiopexy; hymenectomy; esophagogastroduodenoscopy; colonoscopy; tymanoplasty; myringotomy; pilondial cyst excision; pain; anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders; Hernia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard of Care (No VR) Randomization (No Intervention): In the standard of care treatment condition, participants will receive the standard CHLA treatment protocol for IV placement and induction of anesthesia. Current standard of care practices at CHLA for outpatient surgery induction will include the following steps. Children may receive midazolam, parental presence during induction and any other intervention or medication chosen by the HCP. The research team will have no input to the decision regarding the use of any therapy.
- VR Randomization (Experimental): When a child is assigned to the VR condition s/he will have the added component of VR distraction during pre-surgical preparation. Children in the VR condition will interact with an immersive 3D virtual environment presented via a HMD (head-mounted display), a helmet with computer screens for each eye. This study will use two HMDs at two possible time points: (1) Prior to and during IV placement, participants will play using the Oculus Go; (2) Prior to and during anesthesia induction, participants will play using the Mira Prism.
  Interventions: Device: Oculus Go VR; Device: Mira Prism VR

INTERVENTIONS:
Device: Oculus Go VR — The Oculus Go is a standalone headset with built-in speakers that runs independently of a smartphone. Via the Oculus Go, participants will engage with BearBlast (developed by AppliedVR). Throughout the world, plush moles play the role of antagonist, standing in for the nuisance and distraction of pain. The VR game is equipped with a head-tracking system, enabling the player to look around the virtual environment. In addition, there is the option to interact with the VR environment using a tap pad located on the side of the helmet. Therefore, the child will be receiving distraction via 3-D visual and auditory sensory, and tactile feedback, thus supplying a multi-sensory immersive experience. The VR HMD runs independently of a smartphone and has active matrix LCDs with high pixel resolution, creating a bright, vibrant color and a quality image.
  Arms: VR Randomization
Device: Mira Prism VR — The Mira Prism is a portable, augmented reality (AR) HMD powered by iPhone. When paired with the iPhone, the Mira Prism goggles can superimpose computer-generated images on the user's view of the real world. Unlike the full immersion of VR, AR allows users to view the outside world while interacting with digital content. In this study, the patient will interact with Magic Mallet (developed by Miney Moe) until falling asleep during the anesthesia induction process. Magic Mallet is a distraction game designed for pain management and communication during procedures. The game automatically adjusts cognitive load for optimal effect for users. Study team iPhones specifically loaded with Magic Mallet, and without cellular capability, will be used with the Mira Prism.
  Arms: VR Randomization

SUMMARY:
This study aims to test the effectiveness of virtual reality (VR) as a non-pharmaceutical intervention to reduce pain and anxiety in children undergoing various procedures in the Ambulatory Surgery Center (ASC) at CHLA, as measured by self- and proxy-report.

DETAILED DESCRIPTION:
4 million children undergo surgery in the US each year and up to 65% of these children experience significant anxiety and distress before surgery. High anxiety can be traumatic, but it can also lead to postoperative adverse outcomes, such as increased pain and analgesics requirements, delayed hospital discharge, and maladaptive behavioral changes, in children after the surgery. Non-pharmacological intervention, complementary and alternative medicine (CAM) interventions, such as virtual reality, has been shown to decrease anxiety and distress in other medical procedures (e.g., burn care, phlebotomy). Yet to date, no clinical trial has been conducted to examine the effectiveness of virtual reality (VR) to reduce anxiety and distress prior to outpatient surgeries in the operating room setting.

The current study aims to: 1) Determine if VR is more effective than standard care for preventing anxiety, distress, and pain before surgery among children undergoing anesthesia induction, 2) To evaluate healthcare provider's and caregiver's assessment of patient cooperation and caregiver's distress and satisfaction with VR compared to standard of care, and 3) to explore the influence of patient and caregiver characteristics on the effectiveness of VR in preventing pre-operative anxiety and distress and subsequent post-operative outcomes.

Study Population: Children (age 10 - 21 years) and their parents who are scheduled to undergo outpatient surgery, whose health status is American Society of Anesthesiologists (ASA) physical status I-III, and are in the normal range of development are eligible to be in the study.

Study Methodology: The study is a randomized, controlled trial designed to examine the effects of VR on the level of preoperative pain, anxiety and distress of children undergoing surgery.

Statistical Analyses: Univariate Analysis of Variance (ANOVA) will be used to compare differences in primary and secondary outcome variables in VR + standard of care to standard of care only conditions when pre and post-operative measures are available. Univariate ANOVA will be used to compare conditions on post-operative variables. Multiple regression analyses will be used to examine the influence of patient and caregiver variables on patient outcomes in the VR group only.

ELIGIBILITY:
Inclusion Criteria:

* Children who are 10-21 years old
* Children who are English speaking (parents may be Spanish English speaking or Spanish speaking)
* Children who are scheduled to undergo outpatient surgery are eligible to participate in this project.
* Children whose health status is American Society of Anesthesiologists (ASA) physical status I-III will be recruited for this study. ASA status I refers to patients who are normal and healthy with no known systemic disease. ASA status II refers to patients who have mild or well-controlled systemic diseases, such as non-insulin dependent diabetes, upper respiratory conditions, well-controlled asthma or allergies.
* Only children who are in the normal range of development will be recruited for this study. This will be assessed by report from the parents. The rationale for excluding patients with developmental delay is that due to their cognitive impairments, such children react to the stressors of surgery differently than do children without such developmental delay. It is unclear how such children would use the preparation programs and interventions included in this study, and it is likely that their responses on baseline and outcome measures will differ from children of normal developmental parameters.

Exclusion Criteria:

* Children with health status defined by ASA status IV-V will be excluded from this study. ASA status IV refers to patients with an incapacitating systemic disease that is a constant threat to life. ASA status V patients are considered moribund.
* Children who are taking psychotropic medications that affect emotion modulation will be excluded from this study.
* Children with organic brain syndrome, mental retardation, or other known cognitive/neurological disorders
* Children with visual, auditory, or tactile deficits that would interfere with the ability to complete the experimental tasks or use the technological devices
* Children with a history of seizure disorder.
* Children currently sick with flu-like symptoms or experiencing a headache or earache

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 450 (Estimated)
Dates: Start 2015-12-04 (Actual); Primary Completion 2026-12-06 (Estimated); Study Completion 2026-12-06 (Estimated)

PRIMARY OUTCOMES:
VAS anticipatory anxiety measure | Approximately 5 minutes to one hour before procedure
  The VAS anticipatory anxiety measure is a vertical VAS, anchored with 0 at the bottom indicating the least amount and 10 at the top indicating the greatest amount, in response to the instruction to rate "how nervous, afraid, or worried" they were about the upcoming task. The scale also has color cues, graded from yellow at the bottom to dark red at the top, as well as a neutral face at the bottom and a face showing a negative expression at the top. Prior research used the VAS to rate anticipatory anxiety and pain in children.
STAI-C (if elementary or junior high aged), STAI-Y (if in high school or college) | Approximately 5 minutes to one hour before procedure
  The STAIC is a self-administered measure of anxiety in children. It is comprised of separate, self-report scales for measuring two distinct anxiety concepts: state anxiety (A-State) and trait anxiety (A-Trait). The STAI-C distinguishes between a general proneness to anxious behavior rooted in the personality and anxiety as a fleeting emotional state. The instrument consists of two 20-item scales. In the current study, the measure will be used to measure both state and trait anxiety. The STAI is the validated instrument for measuring anxiety in in elementary and junior high aged children.
Child State Anxiety Index (CASI) or Anxiety Sensitivity Index (ASI) if 18 and older | Approximately 5 minutes to one hour before procedure
  The Childhood Anxiety Sensitivity Index (CASI): CASI is an 18-item scale that measures the tendency to view anxiety-related bodily sensations as dangerous (e.g., ''It scares me when my heart beats fast''). Items are scored on a 3-point scale (none, some, a lot), and total scores are calculated by summing all items. The CASI has demonstrated high internal consistency and adequate test-retest reliability. The CASI correlates well with measures of trait anxiety but also accounts for variance in fear not attributable to trait anxiety measures.
The Faces Pain Scale (FPS-R) | Approximately 5 minutes to one hour before procedure
  Revised is an updated version of the Wong-Baker Faces Pain Rating Scale depicting no pain as a neutral expression as compared with the smiling face of the original measure. The child is asked to point to the face cartoon that depicts how they are currently feeling because of their pain. Face measures are thought to measure pain intensity, and the Wong-Baker Faces measure has demonstrated good reliability and validity.
Child Satisfaction Questionnaire | Approximately 5-15 minutes after procedure
  The child survey is 13-item, Likert-like survey to assess child estimates of pain reduction, fear reduction, decreased behavioral distress, and overall satisfaction; it mirrors the parent survey. There are two versions, one for each treatment condition. Two versions of the survey exist, to account for condition (VR vs. standard of care).
CAMPIS-R | Peri-procedure
  The CAMPIS-R is a standardized rating scale that codes videotaped verbal interactions in the pediatric treatment room. The CAMPIS-R codes the subject, speaker, phase of medical procedure, verbal content, affective tone, and to whom vocalizations are directed. Adult vocalizations are coded as coping-promoting (nonprocedural talk or humor directed to the child, commands to engage in coping strategies), distress-promoting (reassuring comments, apologies, giving control to the child, criticism, and empathetic statements), or neutral (humor to adults, nonprocedural talk to adults, child's condition talk, commands for procedural activity, praise, notification of procedure to come, behavioral commands to child, checking child's status).
Yale Preoperative Anxiety Scale (m-YPAS; Kain et al., 1995; Kain et al., 1997) | Peri-procedure
  The YPAS consists of 27 items in five domains of behavior indicating anxiety in young children (Activity, Emotional expressivity, State of arousal, Vocalization and Use of parents). This measure takes approximately 5-10 minutes to complete. The 'adjusted YPAS total score' ranges from 0 to 100 with higher scores indicating greater anxiety. The YPAS was developed originally to measure the anxiety of children while undergoing induction of anesthesia. Recently, we validated the YPAS against a self-report measure, the State Trait Anxiety Inventory for Children (Kain et al., 1997; STAIC). Data Obtained: Standard scores for the anxiety level of children during the perioperative period.
Parent Anxiety Scale | Approximately 5 minutes to one hour before procedure
  The parent is asked to indicate "how nervous, afraid, or worried" they believe their child was about the task on a scale of 1 to 10, from least to most anxious. (See description of Child Anticipatory/Procedural Anxiety)
STAI | Approximately 5 minutes to one hour before procedure
  The STAI is a self-administered measure of anxiety in adults. It is comprised of separate, self-report scales for measuring two distinct anxiety concepts: state anxiety (A-State) and trait anxiety (A-Trait). The STAI-Y distinguishes between a general proneness to anxious behavior rooted in the personality and anxiety as a fleeting emotional state. The instrument consists of two 20-item scales. In the current study, the measure will be used to measure trait and state anxiety. The STAI is the validated instrument for measuring anxiety in working adults, and in young adults in high school and college.
Parent Pain Scale | Approximately 5-15 minutes after procedure
  Parents/Caregivers will be asked to report on their child's pain on a faces pain scale of 1 to 6, from least to most pain, during 1) the IV start procedure and 2) the mask induction. (See description of Child Pain - POST)
7-item self-report measure of healthcare provider's perceptions about the child's cooperation, pain, distress, and anxiety | Peri-procedure
  The healthcare provider survey is a 7-item Likert-like investigator-developed survey to assess their estimates of pain and anxiety management, cooperation, and satisfaction with the procedure. Healthcare providers are also invited to write comments about the use of VR (if applicable) during the IV placement procedure.
6-item self-report measure of healthcare provider's perceptions about the child's cooperation, distress, and anxiety | Peri-procedure
  The healthcare provider survey is a 6-item Likert-like investigator-developed survey to assess their estimates of fear reduction, decreased behavioral distress, and overall satisfaction related to the procedure they just performed with the child/adolescent. Healthcare providers are also asked about sedative use and are invited to write comments about the use of VR (if applicable) during the mask induction procedure.
VAS anticipatory anxiety measure | Approximately 5-15 minutes after procedure
  The VAS anticipatory anxiety measure is a vertical VAS, anchored with 0 at the bottom indicating the least amount and 10 at the top indicating the greatest amount, in response to the instruction to rate "how nervous, afraid, or worried" they were about the upcoming task. The scale also has color cues, graded from yellow at the bottom to dark red at the top, as well as a neutral face at the bottom and a face showing a negative expression at the top. Prior research used the VAS to rate anticipatory anxiety and pain in children.
STAI-C (if elementary or junior high aged), STAI-Y (if in high school or college) | Approximately 5-15 minutes after procedure
  The STAIC is a self-administered measure of anxiety in children. It is comprised of separate, self-report scales for measuring two distinct anxiety concepts: state anxiety (A-State) and trait anxiety (A-Trait). The STAI-C distinguishes between a general proneness to anxious behavior rooted in the personality and anxiety as a fleeting emotional state. The instrument consists of two 20-item scales. In the current study, the measure will be used to measure both state and trait anxiety. The STAI is the validated instrument for measuring anxiety in in elementary and junior high aged children.
The Faces Pain Scale (FPS-R) | Approximately 5-15 minutes after procedure
  Revised is an updated version of the Wong-Baker Faces Pain Rating Scale depicting no pain as a neutral expression as compared with the smiling face of the original measure. The child is asked to point to the face cartoon that depicts how they are currently feeling because of their pain. Face measures are thought to measure pain intensity, and the Wong-Baker Faces measure has demonstrated good reliability and validity.
Parent Anxiety Scale | Approximately 5-15 minutes after procedure
  The parent is asked to indicate "how nervous, afraid, or worried" they believe their child was about the task on a scale of 1 to 10, from least to most anxious. (See description of Child Anticipatory/Procedural Anxiety)
STAI | Approximately 5-15 minutes after procedure
  The STAI is a self-administered measure of anxiety in adults. It is comprised of separate, self-report scales for measuring two distinct anxiety concepts: state anxiety (A-State) and trait anxiety (A-Trait). The STAI-Y distinguishes between a general proneness to anxious behavior rooted in the personality and anxiety as a fleeting emotional state. The instrument consists of two 20-item scales. In the current study, the measure will be used to measure trait and state anxiety. The STAI is the validated instrument for measuring anxiety in working adults, and in young adults in high school and college.

SECONDARY OUTCOMES:
Malaise Scale (MS) | Approximately 5 minutes to one hour before procedure
  The MS is a six-point scale indicating level of nausea from (1) no symptoms to (6) being sick The MS is completed before and after administration of the VR game to monitor for any signs of nausea. Instructions to the child are as follows: "This is a scale from one to six. One means that you feel fine and no different to how you normally feel. Two means that you feel a little bit different or funny but not sick in the tummy. Three means that you feel a little bit sick and four means that you feel more than a little bit sick but not really sick. Five means that you feel really sick, like you are going to throw up or vomit and six means that you are being sick or vomiting. I'm going to ask you every few minutes how you feel. I want you to tell me which number from one to six best describes how you feel at that time."
Blood pressure and heart rate (BP/ HR) | Approximately 5 minutes to one hour before procedure
  Blood pressure and heart rate assessed intraoperatively and in the operating room will be ascertained via chart review.
Child Presence Questionnaire | Approximately 5-15 minutes after procedure
  The Child Presence Questionnaire was developed out of a content analysis of the entire domain of adult presence items and selection and adaptation of appropriate items for assessing the child's sense of believability of their experience. This 16-item measure is verbally administered to children and asks them to respond according to a 3-point Likert-like format. Items assess the child's sense of involvement, realism, and transportation into the experience. Patients in the VR condition will complete the Child Presence Questionnaire post-procedure to assess level of VR immersion.
Behavior Assessment System for Children (BASC-2) | Approximately 5 minutes to one hour before procedure
  The BASC-2 is a multi-dimensional approach to evaluate behavior (problem behavior as well as adaptive behavior) of children 8 to 18 years old. The parent-report measure has good internal consistency and test-retest reliability. It has been validated in English and Spanish.
Parent Satisfaction Questionnaire | Approximately 5-15 minutes after procedure
  The parent survey is 16-item, Likert-like survey to assess parent estimates of pain reduction, fear reduction, decreased behavioral distress, and overall satisfaction. Two versions of the survey exist, to account for condition (VR vs. standard of care).
Pediatric Anesthesia Emergence Delirium (Sikich, 2004; PAED) | Approximately 5-15 minutes after procedure
  The PAED rating scale consists of five psychometric items ("child makes eye contact with the caregiver", "child's actions are purposeful", child is aware of the surroundings", child is restless", "child is inconsolable") for the measurement of ED in children. A decreased ability of the child to make eye contact with the caregiver and a declined awareness of his surroundings reflect disturbances in consciousness with a reduced ability to focus, sustain, or shift attention. Less purposeful actions suggest cognitive changes that include perception and memory impairment as well as disorganized thinking patterns. The two other items reflect a disturbance in psychomotor behavior and emotion, although they may also suggest pain or apprehension.
Watcha Scale (Watcha et al., 1992) | Approximately 5-15 minutes after procedure
  The Watcha Scale is a four point scale that is used to assess emergence delirium (ED). A child with a score of 3 or 4 can be considered to have emergence delirium. The Watcha Scale demonstrates reliability and validity in pediatric populations (Reduque & Verghese 2012).
Analgesic Requirements | Peri-procedure
  Frequency and dose of analgesic administered intraoperatively and in the operating room will be ascertained via chart review. Data Obtained: Frequency and dose of analgesic received in the operating room.
Malaise Scale (MS) | Approximately 5-15 minutes after procedure
  The MS is a six-point scale indicating level of nausea from (1) no symptoms to (6) being sick The MS is completed before and after administration of the VR game to monitor for any signs of nausea. Instructions to the child are as follows: "This is a scale from one to six. One means that you feel fine and no different to how you normally feel. Two means that you feel a little bit different or funny but not sick in the tummy. Three means that you feel a little bit sick and four means that you feel more than a little bit sick but not really sick. Five means that you feel really sick, like you are going to throw up or vomit and six means that you are being sick or vomiting. I'm going to ask you every few minutes how you feel. I want you to tell me which number from one to six best describes how you feel at that time."

OTHER OUTCOMES:
Demographic Survey | Approximately 5 minutes to one hour before procedure
  A brief demographic survey will be administered to parent regarding their child's age, ethnicity, grade in school, and any medical conditions or learning problems they may have.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey I Gold, PhD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perry JN, Hooper VD, Masiongale J. Reduction of preoperative anxiety in pediatric surgery patients using age-appropriate teaching interventions. J Perianesth Nurs. 2012 Apr;27(2):69-81. doi: 10.1016/j.jopan.2012.01.003. PMID 22443919
- [Background] Davidson A, McKenzie I. Distress at induction: prevention and consequences. Curr Opin Anaesthesiol. 2011 Jun;24(3):301-6. doi: 10.1097/ACO.0b013e3283466b27. PMID 21494130
- [Background] Kain ZN, Mayes LC, O'Connor TZ, Cicchetti DV. Preoperative anxiety in children. Predictors and outcomes. Arch Pediatr Adolesc Med. 1996 Dec;150(12):1238-45. doi: 10.1001/archpedi.1996.02170370016002. PMID 8953995
- [Background] Kain Z, Lc M, Cote C, Todres D: The perioperative behavioral stress response in children, Practice of Anesthesia for Infants and Children. Edited by Anonymous. Philadelphia, W.B. Saunders, 2001, pp 25-37.
- [Background] Kain Z, Mayes L, Borestein M, Genevro J: Anxiety in children during the perioperative period, Child Development and Behavioral Pediatrics. Edited by Anonymous. Mahwah, NJ, Lawrence Erlbaum Associates, 1996, pp 85-103.
- [Background] Burton L, Verma V: Anxiety relating to illness and treatment, Anxiety in Children. Edited by Anonymous. New York, Methuen Croom Helm, 1984, pp 151-172.
- [Background] Kain Z, Atlee J: Perioperative psychological trauma in children, Complications in Anesthesiology. Edited by Anonymous. Philadelphia, WB Saunders, 1999, pp 674-677.
- [Background] Kain ZN, Wang SM, Mayes LC, Caramico LA, Hofstadter MB. Distress during the induction of anesthesia and postoperative behavioral outcomes. Anesth Analg. 1999 May;88(5):1042-7. doi: 10.1097/00000539-199905000-00013. PMID 10320165
- [Background] Kain Z, Sevarino F, Rinder C: The preoperative behavioral stress response: Does it exist? Anesthesiology 1999; 91: A742.
- [Background] Kiecolt-Glaser JK, Page GG, Marucha PT, MacCallum RC, Glaser R. Psychological influences on surgical recovery. Perspectives from psychoneuroimmunology. Am Psychol. 1998 Nov;53(11):1209-18. doi: 10.1037//0003-066x.53.11.1209. PMID 9830373
- [Background] Johnston M. Pre-operative emotional states and post-operative recovery. Adv Psychosom Med. 1986;15:1-22. doi: 10.1159/000411845. No abstract available. PMID 3706030
- [Background] Kain ZN, Sevarino F, Alexander GM, Pincus S, Mayes LC. Preoperative anxiety and postoperative pain in women undergoing hysterectomy. A repeated-measures design. J Psychosom Res. 2000 Dec;49(6):417-22. doi: 10.1016/s0022-3999(00)00189-6. PMID 11182434
- [Background] Martinez-Urrutia A. Anxiety and pain in surgical patients. J Consult Clin Psychol. 1975 Aug;43(4):437-42. doi: 10.1037/h0076898. No abstract available. PMID 1159142
- [Background] Wallace LM. Pre-operative state anxiety as a mediator of psychological adjustment to and recovery from surgery. Br J Med Psychol. 1986 Sep;59(3):253-61. doi: 10.1111/j.2044-8341.1986.tb02691.x. PMID 3768273
- [Background] Kain ZN. Premedication and parental presence revisited. Curr Opin Anaesthesiol. 2001 Jun;14(3):331-7. doi: 10.1097/00001503-200106000-00009. PMID 17019112
- [Background] Kain ZN, Caldwell-Andrews AA, LoDolce ME, Krivutza DM, Wang SM: The Perioperative Behavioral Stress Response in Children. Anesthesiology 2002; 96: A1242.
- [Background] Viitanen H, Annila P, Viitanen M, Tarkkila P. Premedication with midazolam delays recovery after ambulatory sevoflurane anesthesia in children. Anesth Analg. 1999 Jul;89(1):75-9. doi: 10.1097/00000539-199907000-00014. PMID 10389782
- [Background] Viitanen H, Annila P, Viitanen M, Yli-Hankala A. Midazolam premedication delays recovery from propofol-induced sevoflurane anesthesia in children 1-3 yr. Can J Anaesth. 1999 Aug;46(8):766-71. doi: 10.1007/BF03013912. PMID 10451136
- [Background] Kain ZN, Caldwell-Andrews AA, Krivutza DM, Weinberg ME, Wang SM, Gaal D. Trends in the practice of parental presence during induction of anesthesia and the use of preoperative sedative premedication in the United States, 1995-2002: results of a follow-up national survey. Anesth Analg. 2004 May;98(5):1252-9, table of contents. doi: 10.1213/01.ane.0000111183.38618.d8. PMID 15105196
- [Background] Chow CH, Van Lieshout RJ, Schmidt LA, Dobson KG, Buckley N. Systematic Review: Audiovisual Interventions for Reducing Preoperative Anxiety in Children Undergoing Elective Surgery. J Pediatr Psychol. 2016 Mar;41(2):182-203. doi: 10.1093/jpepsy/jsv094. Epub 2015 Oct 17. PMID 26476281
- [Background] Hoffman HG, Patterson DR, Carrougher GJ, Sharar SR. Effectiveness of virtual reality-based pain control with multiple treatments. Clin J Pain. 2001 Sep;17(3):229-35. doi: 10.1097/00002508-200109000-00007. PMID 11587113
- [Background] Mahrer NE, Gold JI. The use of virtual reality for pain control: a review. Curr Pain Headache Rep. 2009 Apr;13(2):100-9. doi: 10.1007/s11916-009-0019-8. PMID 19272275
- [Background] Malloy KM, Milling LS. The effectiveness of virtual reality distraction for pain reduction: a systematic review. Clin Psychol Rev. 2010 Dec;30(8):1011-8. doi: 10.1016/j.cpr.2010.07.001. Epub 2010 Jul 13. PMID 20691523
- [Background] Reger, G. M., A. A. Rizzo, J. G. Buckwalter, J. Gold, R. Allen, R. Augustine, and E. Mendelowitz.
- [Background] Gold JI, Kim SH, Kant AJ, Joseph MH, Rizzo AS. Effectiveness of virtual reality for pediatric pain distraction during i.v. placement. Cyberpsychol Behav. 2006 Apr;9(2):207-12. doi: 10.1089/cpb.2006.9.207. PMID 16640481
- [Background] Jeffs D, Dorman D, Brown S, Files A, Graves T, Kirk E, Meredith-Neve S, Sanders J, White B, Swearingen CJ. Effect of virtual reality on adolescent pain during burn wound care. J Burn Care Res. 2014 Sep-Oct;35(5):395-408. doi: 10.1097/BCR.0000000000000019. PMID 24823326
- [Background] Faber AW, Patterson DR, Bremer M. Repeated use of immersive virtual reality therapy to control pain during wound dressing changes in pediatric and adult burn patients. J Burn Care Res. 2013 Sep-Oct;34(5):563-8. doi: 10.1097/BCR.0b013e3182777904. PMID 23970314
- [Background] Kipping B, Rodger S, Miller K, Kimble RM. Virtual reality for acute pain reduction in adolescents undergoing burn wound care: a prospective randomized controlled trial. Burns. 2012 Aug;38(5):650-7. doi: 10.1016/j.burns.2011.11.010. Epub 2012 Feb 18. PMID 22348801
- [Background] Schneider SM, Workman ML. Effects of virtual reality on symptom distress in children receiving chemotherapy. Cyberpsychol Behav. 1999;2(2):125-34. doi: 10.1089/cpb.1999.2.125. PMID 19178248
- [Background] Sinha M, Christopher NC, Fenn R, Reeves L. Evaluation of nonpharmacologic methods of pain and anxiety management for laceration repair in the pediatric emergency department. Pediatrics. 2006 Apr;117(4):1162-8. doi: 10.1542/peds.2005-1100. PMID 16585311
- [Background] Mosso-Vazquez JL, Gao K, Wiederhold BK, Wiederhold MD. Virtual reality for pain management in cardiac surgery. Cyberpsychol Behav Soc Netw. 2014 Jun;17(6):371-8. doi: 10.1089/cyber.2014.0198. PMID 24892200
- [Background] Dahlquist LM, Weiss KE, Clendaniel LD, Law EF, Ackerman CS, McKenna KD. Effects of videogame distraction using a virtual reality type head-mounted display helmet on cold pressor pain in children. J Pediatr Psychol. 2009 Jun;34(5):574-84. doi: 10.1093/jpepsy/jsn023. Epub 2008 Mar 26. PMID 18367495
- [Background] Dahlquist LM, McKenna KD, Jones KK, Dillinger L, Weiss KE, Ackerman CS. Active and passive distraction using a head-mounted display helmet: effects on cold pressor pain in children. Health Psychol. 2007 Nov;26(6):794-801. doi: 10.1037/0278-6133.26.6.794. PMID 18020853